CLINICAL TRIAL: NCT04266483
Title: Cancer Genome Atlas of China:Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: ChosenMed Technology (Beijing) Co.,Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: YCZYPT[2018]06-01
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Next-generation sequencing; High-throughput sequencing; Gene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 10ml anticoagulant peripheral blood and lung cancer tumor tissue which should meet one of the following requirements: fresh tissue samples (more than 1cm, at least 2 pieces) obtained by operation (1 piece， soybean size) or needle biopsy , 2 pieces of bronchoscopic biopsy tissue, paraffin section (thickness between 4 to 8 μ m, operation or biopsy samples, more than 10 pieces, unstained)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on 2500 lung cancer tumor tissue samples from about 40 clinical centers in China, the molecular typing of lung cancer in China will be figured out by high throughput sequencing, which will provide the basis for the follow-up research and development of new drugs as well as the guidance of treatment.

DETAILED DESCRIPTION:
This project will establish a standardized procedure of lung cancer sample collection, transportation, storage, detection, bioinformatics analysis and result judgment, so as to draw up the gene map of advanced lung cancer in China, and provide an important basis for the research and development of new drugs and the guidance of treatment.

Firstly, 2500 cases of lung cancer tumor tissue samples will be collected according to the Inclusion Criteria.

Secondly，samples will be sequenced through high throughput sequencing by ChosenMed Technology (Beijing) Co., Ltd., according to the strict process. Panel sequencing of the samples will be carried out through Illumina platform. After targeting Panel sequencing, four types of mutations including point mutation, insertion deletion, gene fusion and copy number variation will be detected, and tumor mutation burden as well as microsatellite instability will be evaluated. Combined with the bioinformatics analysis and sequencing results of the samples, the gene map of lung cancer in China will be drawn up, and the specific multigene panel of lung cancer for the Chinese population will be established as the basis for the subsequent clinical screening of molecular markers related to targeting therapy, immunotherapy and prognosis.

Thirdly, patients will be followed up on the information related to treatment after sequencing. According to the genetic information of the patients, the curative effect and prognosis of the patients will be followed up every three to six months. The follow-up time includes at least the first treatment plan after the patients' detection, which may continue until the final survival time of the patients, and explore the molecular markers and combinations that can affect the curative effect and prognosis of patients with lung cancer.

Finally, the clinical data and specimen information of patients will be managed and analyzed by Excel. Multivariate Cox regression analysis will be used to explore the clinical, pathological and molecular markers that affect the prognosis and curative effect of lung cancer, and draw the survival curve with the statistically significant indicators so as to provide reliable statistical results for the following clinical guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed advanced non-small cell lung cancer
2. Stage Ⅲ or Ⅳ non-small cell lung cancer and should to receive tyrosine kinase inhibitors or immune checkpoint inhibitors for the first-line or adjuvant treatment
3. Able to provide 10ml anticoagulant peripheral blood and tumor tissue which should meet at least one of the following requirements: fresh tissue samples (≥ 1cm, at least 2 pieces) obtained by operation (1 piece, soybean size) or needle biopsy, 2 pieces of bronchoscopic biopsy tissue, paraffin section (thickness of 4-8 μm, operation or biopsy samples, ≥ 10 pieces, unstained)
4. Able to provide basic clinical and pathological data
5. Must be willing to be followed up

Exclusion Criteria:

1. Small cell lung cancer
2. Stage I or II non-small cell lung cancer
3. Be not able to provide enough peripheral blood or tumor tissue
4. Incomplete basic clinical data
5. Unwilling to be followed up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage Ⅲ or Ⅳ non-small cell lung cancer who are to receive tyrosine kinase inhibitors or immune checkpoint inhibitors for the first-line or adjuvant treatment.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-11-08 (Estimated); Study Completion 2022-11-08 (Estimated)

PRIMARY OUTCOMES:
Predictive gene profiles | Follow up at least three years
  Concordance between specific gene profiles and treatment outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Xiuyi Zhi, M.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (31):
- China (31):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou Institute of Respiratory Health, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Jilin University, Changchun, Jilin
  - Sino-Japan Friendship Hospital, Jilin University, Changchun, Jilin
  - The Third Hospital of Jilin University, Changchun, Jilin
  - The First Hospital Affiliated to Dalian Medical University, Dalian, Liaoning
  - General Hospital of the Northern Theater of Chinese PLA, Shenyang, Liaoning
  - The First Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shangdong
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine (Binjiang District), Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medcine (Headquarters), Hangzhou, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - The Fourth Medical Center of PLA General Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital,Beijing, Beijing
  - Air Force Specialized Medical Center, Beijing
  - Peking University Cancer Hospital, Beijing
  - The Seventh Medical Center of PLA General Hospital, Beijing
  - Beijing Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Renji Hospital,Shanghai Jiaotong University School of Medicine, Shanghai
  - Lung Hospital Affiliated to Shanghai Tongji Medical University, Shanghai
  - General Hospital of Tianjin Medical University, Tianjin

IPD SHARING:
Plan to Share IPD: No